CLINICAL TRIAL: NCT06229418
Title: Developing and Testing Drone-Delivered AEDs for Cardiac Arrests In Rural America
Acronym: RESTORe-CARE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Virginia Commonwealth University (Other); University of Toronto (Other); University of Washington (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro00113925; 23HERNPRH1150361 (Other Grant/Funding Number: AHA)
Record Dates: First submitted 2024-01-19; First posted 2024-01-29 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-07

CONDITIONS: Cardiac Arrest; Sudden Cardiac Arrest
Keywords: Drone; Automated External Defibrillator
MeSH Terms: conditions — Heart Arrest; Death, Sudden, Cardiac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DFR AED Program (Experimental): Real-time and simulated out-of-hospital cardiac arrests that occur across 6 communities (4 rural, 2 urban)
  Interventions: Other: DFR AED Pilot Program

INTERVENTIONS:
Other: DFR AED Pilot Program — Integrate AED drone delivery into an existing FAA-approved drone-as-first-responder programs

SUMMARY:
The overall goal of this project is to design, develop, and pilot test an emergency healthcare drone delivery system suitable for rural communities that can deliver AEDs to out-of-hospital cardiac arrest (OHCA) locations more rapidly than can be achieved with current first responder and EMS systems. The goal is to determine whether this method of AED delivery can be achieved rapidly enough to justify a future clinical trial directly testing its ability to improve OHCA survival.

DETAILED DESCRIPTION:
To achieve the project goal, 3 specific aims will be addressed. The details in this ClinicalTrials.gov record are specific to Aim 3.

Aim 1:

Define options for emergency healthcare drone station configurations best suited for rural communities and use these findings to help design future drone AED delivery programs in rural communities.

Sub aim 1a:

Define and examine EMS agency treatment, performance, and outcomes of OCHA in rural versus urban regions across the US. This will be done by using CARES Registry data from all OHCA treated by emergency medical professionals from participating EMS agencies in the US between 2021-2022.

Sub aim 1b:

Develop an optimization model to examine the effectiveness of different options for placement of both public and drone-delivered AEDs in rural communities. This will be done by using CARES Registry data from OHCAs between 2012-2022 from participating EMS agencies in North Carolina.

Aim 2:

Develop procedural and operational infrastructure for drone AED delivery that can be applied to rural communities. The primary objective of this aim will be to demonstrate that drone AED delivery can be integrated effectively into existing FAA-approved drone-as-first responder programs.

Aim 3:

Pilot test the safety and effectiveness of emergency drone AED delivery models in 2 urban and 4 rural communities in Forsyth County, NC and James City County, VA.

Sub aim 3a:

Test the ability of the DRF-AED program to travel to the location of suspected OHCAs and arrive ahead of EMS. There will be 12-15 OHCAs across the 6 communities during this testing period.

Sub aim 3b:

Test the ability of the DRF-AED program to deliver and safely deploy AEDs (without interrupting bystanders) to sites of suspected OHCA. There will be 10-12 (with a maximum of 15) additional OCHAs across the 6 communities.

Sub aim 3c:

Test the ability of the DRF-AED program to deliver an AED and treat an OCHA patient suspected cardiac arrests. Up to 70 OHCAs are expected across all 6 communities.

Sub aim 3d:

Carry out simulated OHCA alerts and test the ability of the DRF-AED program to deliver AEDs to a simulated OCHA scene ahead of EMS or first responders. A minimum of 40 simulations of OHCA (10 per rural community) to occur.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age or older in the CARES registry who suffer cardiac arrest before arrival of a 911-responder of non-traumatic cause, including patients who receive an AED shock by a bystander prior to the arrival of 911 responders.

Exclusion Criteria:

* Patients in the CARES registry who have a traumatic cause of cardiac arrest.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2025-12-31 (Estimated); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Time interval difference between AED arrival of drones versus law/fire/EMS arrival to the OCHA scene | 6 months (Aim 3a)
Time interval difference between AED arrival of drones versus law/fire/EMS arrival to the OCHA scene | 15 months (Aim 3c)

SECONDARY OUTCOMES:
Proportion of OHCA cases with drone arrival ahead of EMS arrival | 6 months (Aim 3a)
Proportion of OHCA cases with drone arrival ahead of EMS arrival | 15 months (Aim 3c)
Proportion of times AED was successfully deployed | 6 months (Aim 3b)
Time from drone arrival on scene to AED delivery on the ground | 6 months (Aim 3b)
Drone altitude at time of deployment | 6 months (Aim 3b)
Rates of bystander AED application | 15 months (Aim 3c)
Proportions of initial shockable rhythm | 15 months (Aim 3c)
Proportion of bystander defibrillation | 15 months (Aim 3c)
Proportion of first responder defibrillation | 15 months (Aim 3c)

CONTACTS AND LOCATIONS:
Overall Officials: Monique Starks, MD, Principal Investigator — Duke University; Daniel Mark, MD, Principal Investigator — Duke University; Joseph Ornato, MD, Principal Investigator — Virginia Commonwealth University

IPD SHARING:
Plan to Share IPD: No